CLINICAL TRIAL: NCT04652557
Title: Randomized Placebo-controlled Phase II Cross-over Study on the Influence of Fampridine on Working Memory in Healthy Subjects
Brief Title: Influence of Fampridine on Working Memory in Healthy Young Subjects
Acronym: FamH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-02828
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Working Memory
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fampridine SR (Experimental): Active study medication consists of 7 tablets of fampridine SR 10 mg formulated for oral administration taken in the morning and evening 12 h apart without food. Tablets must be administered whole.
  There will be a washout period of at least 8 days equaling over 30 half-lives of the active substance fampridine (t½ = 6 h) between experimental and control intervention and up to 82 days depending on the individual scheduling of each subject.
  Interventions: Drug: Fampridine SR
- Placebo (Placebo Comparator): Identically looking placebo tablets consisting of widely identical additives formulated for oral administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fampridine SR — Fampridine SR is an inhibitor of voltage gated potassium channels and is approved in Switzerland for treatment of gait problems in patients with Multiple Sclerosis (MS).
  Arms: Fampridine SR
Drug: Placebo — no active component
  Arms: Placebo

SUMMARY:
Proof of concept study on the acute effects on working memory of 10 mg fampridine SR as well as the effects after repeated administration of 10 mg twice daily (3.5 days).

The hypothesis ist that fampridine improves working memory performance.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* generally healthy
* normotensive (BP between 90/60mmHg and 140/90mmHg)
* BMI between 19 and 29,9 kg/m2
* aged between 18 and 30 years
* fluent German-speaking
* IC as documented by signature
* at least double vaccination against Covid-19

Exclusion criteria:

* contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to 4-aminopyridine
* use of potassium channel blockers within the last 3 months
* concomitant treatment with OCT 2 inhibitors and substrates (e.g. cimetidine, propranolol)
* acute or chronic psychiatric disorder (e.g. major depression, psychoses, somatoform disorder, suicidal tendency)
* acute cerebrovascular condition
* history of seizures
* risk of lowered seizure threshold (due to e.g. sleep deprivation, withdrawal of alcohol after alcohol abuse)
* renal impairment
* history of malignant cancers
* walking problems (e.g. due to dizziness)
* bradycardia > 50/min during clinical examination
* clinically significant concomitant disease states (e.g. hepatic dysfunction, cardiovascular disease, diabetes, asthma)
* clinically significant laboratory or ECG abnormality that could be a safety issue in the study
* known or suspected non-compliance
* drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language or psychological problems of the participant
* participation in another study with an investigational drug within the 30 days preceding and during the present study
* prior participation (less than two years ago) in a study investigating working memory (notably the n-back task)
* enrolment of the investigator, his/her family members, employees and other dependent persons
* smoking (>3 cigarettes per day)
* intake of psychoactive drugs (e.g. benzodiazepines, antidepressants, neuroleptics)
* pregnancy or breast feeding
* experiencing a syncope during basal rMT measuring
* metal in the brain, skull or elsewhere in the body (e.g., splinters, fragments, clips, etc.)
* implanted neurostimulator (e.g., DBS, epidural/subdural, VNS)
* cardiac pacemaker or intracardiac lines
* medication infusion device
* piercings, pivot teeth (retainers are no exclusion criterion)
* tattoos (head area) less than 3 months old or older than 20 years
* condition after neurosurgery
* hearing problems or tinnitus
* not able to sit still due to tremor, tics, itching
* history of repeated syncope
* head trauma diagnosed as concussion or associated with loss of consciousness
* diagnosis of epilepsy, or a convulsion or a seizure in the past of the participant or his family
* TMS in the past showing problems
* MRI in the past showing problems
* surgical procedures to spinal cord
* spinal or ventricular derivations

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
High-load working-memory performance after repeated administrations (3.5 days) | test days 2 and 4 (end of treatment periods; 4 hours after last intake of fampridine SR) to assess changes between the Verum and Placebo condition
  It will be used the letter n-back task (Heck, Fastenrath et al. 2014)) which includes a 3-back task assessing working memory. The 3-back task requires participants to respond to a letter repeat with two intervening letters (for example, S-m-b-s-g…). Performance will be quantified with the d' measure controlling for false positives. It will be used parallel versions (different sequences) for the four test days. Primary outcome will be performance after repeated intake of study medication.

SECONDARY OUTCOMES:
High-load working-memory performance after acute administration | test days 1 and 3 (beginning of treatment periods; 4 hours after first intake of fampridine SR) to assess differences between the Verum and Placebo condition
  It will be used the letter n-back task (Heck, Fastenrath et al. 2014)) which includes a 3-back task assessing working memory. The 3-back task requires participants to respond to a letter repeat with two intervening letters (for example, S-m-b-s-g…). Performance will be quantified with the d' measure controlling for false positives. It will be administered parallel versions (different sequences) for the four test days. Primary outcome will be performance after repeated intake of study medication.
Reaction time after acute and repeated intake | test days 1 and 3 (beginning of treatment periods; 4 hours after first intake of fampridine SR) to assess differences between the Verum and Placebo condition
  Reaction time for correct answers in the 3-back (d') task (see outcomes 1 and 2)
Attention after acute and repeated administration | first and last day of treatment periods (each 4 hours after intake in the morning); to assess differences between the Verum and Placebo condition
  Performance in a 0-back task (d' measure controlled). It will be used parallel versions (different sequences) for the four test days.
Symbol Digit Modalities Test (SDMT; Smith 1973) after acute and repeated intake | first and last day of treatment periods (each 4 hours after intake in the morning); to assess differences between the Verum and Placebo condition
  The test consists of the presentation of a series of 9 symbols, each of them is paired with a single digit, labeled 1-9, in a key at the top of a sheet. The remainder of the page has a pseudo-randomized sequence of the symbols and the participant must respond with the digit associated with each of these as quickly as possible. The score is the number of correct answers in 90 seconds (max. 110). The administration of SDMT will be preceded by a learning sequence at both timepoints. It will be used parallel versions for all test days.
Fluid intelligence (Gf): Bochumer Matrizentest (BOMAT) | first and last day of treatment periods (each 4 hours after intake in the morning); to assess differences between the Verum and Placebo condition
  Bochumer Matrizentest (BOMAT - advanced -short; Hossiep/Turck/Hasella, 2001, 1st edition), matrix reasoning. It will be administered the BOMAT to measure fluid intelligence (Gf) consisting of 20 items (maximum 20 correct answers possible). Parallel versions will be used for the four test days. It will be used a time-limited version according to Jaeggi (Jaeggi 2010).
Working-memory: Digit Span Task | first and last day of treatment periods (each 4 hours after intake in the morning); to assess differences between the Verum and Placebo condition
  Working memory will be also assessed with the digit span task, a subtest of the "Wechsler Intelligenztest für Erwachsene" (WIE;(von Aster 2006)). Total scores for digit span forward and backward will be calculated as described in the manual of the WIE. Parallel version will be used for the four test days.
Resting motor threshold (rMT) | test days 2 and 4 (last day of treatment periods; approx. 5 hours after last intake of fampridine SR) to assess differences between the Verum and Placebo condition
  The resting motor threshold (rMT) will be measured by transcranial magnetic stimulation (TMS). rMT will be determined by measuring the motor evoked potential (MEP) in the abductor digiti minimi according to Rossini (2001). rMT will be defined as the lowest stimulation intensity by stimulating the primary motor cortex of the left or right hemisphere required to induce an MEP in the abductor digiti minimi of the dominant hand in at least 5 out of 10 trials.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Chair — University of Basel, Transfaculty Research Platform; Andreas Papassotiropoulos, Prof. MD, Study Chair — University of Basel, Transfaculty Research Platform
Locations (1):
- University of Basel, Transfaculty Research Platform, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underline results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available after publication, study protocol (including statistical analysis plan) will be made available before start of the study.
Access Criteria: All IPD (de-identified) that underline results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Request will be reviewed by the team of the principal investigator.

REFERENCES:
- [Derived] Papassotiropoulos A, Freytag V, Schicktanz N, Gerhards C, Aerni A, Faludi T, Amini E, Muggler E, Harings-Kaim A, Schlitt T, de Quervain DJ. The effect of fampridine on working memory: a randomized controlled trial based on a genome-guided repurposing approach. Mol Psychiatry. 2025 May;30(5):2085-2094. doi: 10.1038/s41380-024-02820-1. Epub 2024 Nov 8. PMID 39516710

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04652557/Prot_SAP_001.pdf